CLINICAL TRIAL: NCT07159620
Title: A Prospective Single-Arm Clinical Study of Venetoclax Combined With Azacitidine, Chidamide, Vindesine, and Dexamethasone in Newly Diagnosed ETP-ALL Like Patients
Brief Title: Venetoclax Combined With Azacitidine, Chidamide, Vindesine, and Dexamethasone in Newly Diagnosed ETP-ALL Like Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025662
Record Dates: First submitted 2025-08-26; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Adult T-cell Leukemia/Lymphoma
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — venetoclax; Azacitidine; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Vindesine; Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Venetoclax Combined with Azacitidine, Chidamide, Vindesine, and Dexamethasone (Experimental): Induction Therapy Phase:
  VACVP induction:Venetoclax: 100mg, d1, 200mg, d2, 400mg, d3-d21, orally. Azacitidine,75mg/m²/day, d1-d7, subcutaneously. Chidamide,10mg, d1-d7, orally. Vindesine, 4mg, d1, intravenous infusion. Dexamethasone,9mg/m²/day, d1-d14; reduced by half on d15-d17; further reduced by half on d18-d21, intravenous infusion or orally.
  Consolidation therapy:
  1. alternate use of HD-MTX-Ara C and VACVP
  2. allogeneic hematopoietic stem cell transplantation (HSCT)
  Interventions: Drug: VEN (Venetoclax); Drug: Azacitidine (AZA); Drug: Chidamide; Drug: vindesine; Drug: Dexamethasone

INTERVENTIONS:
Drug: VEN (Venetoclax) — Orally
Drug: Azacitidine (AZA) — Subcutaneous injection
Drug: Chidamide — Orally
Drug: vindesine — intravenous infusion
Drug: Dexamethasone — intravenous infusion or orally

SUMMARY:
ETP-ALL like patients have poor outcomes and prognosis, and the optimal therapeutic approaches are poorly characterized. The goal of this clinical trial is to evaluate the efficacy and safety of the venetoclax combined with azacitidine, chidamide, vindesine, and dexamethasone regimen in newly diagnosed ETP-ALL like patinets (including ETP-ALL, near ETP-ALL and T-ALL with myeloid mutations) .

ELIGIBILITY:
Inclusion Criteria:

1. Age: >14 to 65 years (inclusive).
2. Diagnosis: Patients diagnosed with ETP-ALL like disease meeting the following flow cytometry immunophenotypic criteria:

   ETP-ALL: CD7+, CD1a-, CD8-, CD5 positivity rate ≤75%, and positive for at least one myeloid/stem cell antigen marker (including but not limited to CD34, CD117, HLA-DR, CD13, CD33, CD11b, or CD65); MPO negative.

   Near-ETP-ALL: CD7+, CD1a-, CD8-, CD5 positivity rate >75%, AND positive for at least one myeloid/stem cell antigen marker (including but not limited to CD34, CD117, HLA-DR, CD13, CD33, CD11b, or CD65); MPO negative.

   T-ALL with myeloid mutations: FLT3, DNMT3A, STAG2, IDH1/IDH2, RUNX1, EZH2, WT1, ASXL1/ASXL2, SF3B1, TET2, BCOR, BCORL1.
3. Newly diagnosed patients who have not received any prior induction therapy before enrollment (excluding hydroxyurea, dexamethasone, low-dose cytarabine, venetoclax with a cumulative dose <0.5g, and leukapheresis).
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2.
5. Expected survival >6 months.
6. Demonstrated capacity to understand the study and willingness to provide informed consent.

Exclusion Criteria:

1. Pregnancy, breastfeeding, or unwillingness to use contraception in women of childbearing potential
2. Presence of uncontrolled active infection (including bacterial, fungal, or viral infections); concurrent active HBV, HCV, or HIV infection.
3. Severe Organ Dysfunction:

   Cardiac Insufficiency: Left ventricular ejection fraction (LVEF) ≤40%, OR history of congestive heart failure, unstable coronary artery disease, or severe arrhythmia.

   Respiratory Failure: Partial pressure of arterial oxygen (PaO₂) ≤60 mmHg. Hepatic Impairment: Total bilirubin ≥2 times the upper limit of normal (ULN), OR alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥3 times ULN.

   Renal Impairment: Serum creatinine ≥2 mg/dL, OR creatinine clearance ≤30 mL/min/1.73m².

   Hypersensitivity: History of hypersensitivity to any of the study drugs or compounds of similar chemical structure.
4. Presence of central nervous system (CNS) leukemia.
5. Any other condition deemed by the investigator to make the subject unsuitable for participation in this trial.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Composite Complete Remission Rate（CRc） after induction therapy | Time from the completion of induction and before consolidation therapy（up to 42 days）
  Rates of complete remission (CR), and complete remission with incomplete hematologic recovery (CRi)

SECONDARY OUTCOMES:
Overall survival（OS） | 2 years
  Time from the date of enrollment to death from any cause or the last follow-up
Relapse-Free Survival(RFS) | 2 years
  The duration from the date of the first complete remisson to the occurrence of relapse, death from any cause, or the last follow-up.
duration of remission (DOR) | 2 years
  Time between the first remission and relapse
AE | Within 30 days after the last chemotherapy
  Adverse events during the chemotherapy treatment.
MRD | At the end of induction（up to 42 days）, 1 cycle of consolidation（up to 42 days）, 2 cycle of consolidation （up to 42 days）and the end of consolidation（up to 42 days）
  Percentage of participants who converted to MRD < 10^-4 by flow cytometry

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided